CLINICAL TRIAL: NCT06545916
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Phase 2 Study to Evaluate Impact of Sunobinop (V117957) on Alcohol Consumption in Subjects Diagnosed With Moderate to Severe Alcohol Use Disorder and Seeking Treatment
Brief Title: Study of Sunobinop on Alcohol Consumption in Alcohol Use Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Imbrium Therapeutics (Industry)
Collaborators: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SUN2003A; 2024-517105-85-00 (EU CTIS Number)
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol consumption; Moderate to severe alcohol use disorder
MeSH Terms: conditions — Alcoholism; Alcohol Drinking

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sunobinop (Experimental)
  Interventions: Drug: Sunobinop
- Placebo to match sunobinop (Placebo Comparator)
  Interventions: Drug: Placebo to match sunobinop

INTERVENTIONS:
Drug: Sunobinop — 1 tablet taken orally at bedtime
  Other Names: V117957
  Arms: Sunobinop
Drug: Placebo to match sunobinop — 1 tablet taken orally at bedtime
  Arms: Placebo to match sunobinop

SUMMARY:
The purpose of this study is to evaluate the efficacy of sunobinop compared to placebo on alcohol consumption in subjects with alcohol use disorder.

ELIGIBILITY:
Key Inclusion Criteria include:

* Male and female age ≥18 years.
* Diagnosis of moderate or severe alcohol use disorder.
* Currently seeking treatment for alcohol use disorder.
* Has 4 or more heavy drinking days (HDD) in each of the 4 weeks prior to baseline visit.

Key Exclusion Criteria include:

* Subjects that meet current DSM-5 criteria for moderate or severe substance use disorder other than alcohol and nicotine.

Other protocol-specific inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Percent heavy drinking days (HDD) | Day 57

SECONDARY OUTCOMES:
Number of standard unit drinks | Day 57
Percent of drinking days (PDD) | Day 57

CONTACTS AND LOCATIONS:
Locations (7):
- United States (4):
  - Belmont Medical Office, Brooklyn, New York
  - Ohio Clinical Trials, Columbus, Ohio
  - Inquest Clinical Research, Baytown, Texas
  - Cebis Usa, Llc, Houston, Texas
- Romania (3):
  - Bio Terra Med SRL, Bucharest
  - Spitalul Universitar De Urgenta Militar Central "Dr. Carol Davila", Bucharest
  - Cabinet Medical Individual Dr. Andreea Popa, Bucharest

IPD SHARING:
Plan to Share IPD: No